CLINICAL TRIAL: NCT04288635
Title: Impact of Metabolite Supplementation to Restore Mitochondrial Dysfunction During Septic Shock: a Preclinical Study: MEFDASE Study
Brief Title: Impact of Metabolite Supplementation to Restore Mitochondrial Dysfunction During Septic Shock: a Preclinical Study
Acronym: MEFDASE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC19_0189
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock; Multiple Organ Failure
Keywords: mitochondrial dysfunction
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Whole blood sample for mitochondrial metabolic assessment, DNA extraction for biogenesis and autophagy genes implication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock admitted in Angers' ICU: Patients aged more than 18, admitted in University Hospital of Angers, who meet the full criteria of septic shock
  Interventions: Biological: Whole blood samples

INTERVENTIONS:
Biological: Whole blood samples — Whole blood samples at admission, from day one to three after admission

SUMMARY:
Septic shock is defined as a subset of sepsis with severe metabolism alterations, leading to organ failure. Septic shock is associated with a high mortality, around 40% according to the SEPSIS 3 definition.

Metabolic alterations are responsible for lactic acidosis, and results in mitochondrial dysfunction.

This study aims at evaluate the impact of exogenous metabolites on restoring mitochondrial function in septic shock patients with lactate acidosis.

Mitochondrial metabolism (quantitative analysis, mitochondrial function) in intact Peripheral Blood Mononuclear Cells (PBMC) will be isolate and analyse from patients at the early phase of septic shock (admission), at day 2 and 4. Participant's medical history will be recorded: renal and liver metabolism, severity scores and outcomes and the need for supportive care in the intensive care unit (ICU) until 28 days after admission.

Furthermore, the investigators will evaluate wether selected metabolites added to the cell culture medium may improve mitochondrial metabolism.

DETAILED DESCRIPTION:
In this prospective study, the investigators will include patients admitted to the medical ICU of Angers University Hospital and meeting the SEPSIS-3 criteria for the definition of septic shock (Sequential Organ Failure Assessment (SOFA) score > 2, hyperlactatemia > 2 mmol/L and sepsis).

Blood samples will be collected during the usual care of initial resuscitation and analyzed in the laboratory INSERM (Institut national de la santé et de la recherche médicale) U1232 (University Hospital of Angers).

Mitochondrial metabolism will be analyzed in freshly isolated PBMC and after culture for 1-3 days, with or without the addition of selected metabolites to the cell culture medium.

The evolution of ketogenesis, mitochondrial function, acidobasic status will be assessed across the time (blood samples at day 2 and 4).

Survival, renal and liver metabolism, severity scores and outcomes and the need for supportive care in the intensive care unit (ICU) until 28 days after admission will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or more
* Patients with criteria for septic shock according to SEPSIS 3 definition (presumed sepsis, with persisting hypotension requiring vasopressors to maintain mean arterial pressure > 65 mmHg and having a serum lactate > 2 mmol/L despite adequate fluid expansion).
* Admitted in the ICU of Angers University Hospital

Exclusion Criteria:

* Minor patients (aged less 18)
* Patient subject to legal protection measures
* Refusal of the patient or his family
* Preexisting mitochondrial disease
* Patient with aplasia
* Pregnant or parturient women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 or more who meet the SEPSIS-3 criteria for septic shock : a presumed sepsis, with persisting hypotension requiring vasopressors to maintain mean arterial pressure > 65 mmHg and having a serum lactate > 2 mmol/L despite adequate fluid expansion, admitted to the medical ICU of Angers University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial metabolism (mitochondrial membrane depolarization and respiration) with the supplementation of metabolite in the cell culture medium | Day 0 (whole blood after cells separation), Day 1-3 after cell culture
  Using Fluorescence-activated cell sorting system to assess the membrane depolarization of the mitochondria and Oroboros system for mitochondrial respiration

SECONDARY OUTCOMES:
Overall survival at 28 days | Day 28
  Survival of patients after ICU admission
Change in organs failure | From Day 0 to Day 4
  Using the Sequential Organ Failure Assessment Score
Change and correlation between lactic acidosis, ketogenesis and mitochondrial function evolutions | From Day 1 to Day 3
  biochemical analysis of blood samples, assessment of mitochondrial metabolism (quantitative and qualitative analysis).
Need for renal replacement therapy during the ICU stay | From Day 1 to Day 28
  Need for renal replacement therapy and its duration
Need for vasopressors during the ICU stay | From Day 1 to Day 28
  Need for vasopressors during the ICU stay and its duration
Need for mechanical ventilation during the ICU stay | From Day 1 to Day 28
  Need for mechanical ventilation during the ICU stay and its duration

CONTACTS AND LOCATIONS:
Overall Officials: Julien DEMISELLE, MD, Principal Investigator — University Hospital of Angers
Locations (1):
- CHU, Angers, Maine et Loire, France

IPD SHARING:
Plan to Share IPD: No